CLINICAL TRIAL: NCT04196179
Title: A Phase 1, Randomized, Double-Blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Determine the Safety, Tolerability, Pharmacokinetics, and Food Effect of ANG-3070 in Healthy Adult Participants
Brief Title: ANG-3070 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angion Biomedica Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ANG-3070-001
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SAD (Experimental): A1 Day 1 ANG-3070 50 mg (n=6) / Placebo (n=2) Oral
  A2 Day 1 ANG-3070 100 mg (n=6) / Placebo (n=2) Oral
  A3 Day 1 ANG-3070 200 mg (n=6) / Placebo (n=2) Oral
  Day 15 ANG-3070 200mg (n=6) / Placebo (n=2) Oral
  A4 Day 1 ANG-3070 400 mg (n=6) / Placebo (n=2) Oral
  A5 Day 1 ANG-3070 600 mg (n=6) / Placebo (n=2) Oral
  D1 Single Dose Food Effect: Day 1 ANG 3070 600 mg *with and without food* (n=6)/ Placebo (n=2) Oral
  Interventions: Drug: ANG3070; Drug: Placebo oral capsule
- MAD (Experimental): B1 ANG-3070 50 mg BID (n=6) / Placebo (n=2)
  B2 ANG-3070 100 mg BID (n=6) / Placebo (n=2)
  B3 ANG-3070 250 mg BID (n=6) / Placebo (n=2)
  B4 ANG-3070 500 mg, BID (n=6)/ Placebo (n=2)
  C1 ANG-3070 400 mg, QD(n=6)/ Placebo (n=2)
  C2 ANG-3070 600 mg, QD (n=6)/ Placebo (n=2)
  Interventions: Drug: ANG3070; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ANG3070 — ANG-3070 drug product is a an immediate release oral solid. The drug product consists of a Size 00 Swedish orange capsule containing drug substance (10 mg, 50 mg, or 250 mg) with no excipients.
Drug: Placebo oral capsule — ANG-3070 placebo capsules visually match the drug product.

SUMMARY:
This is a Phase 1 study, to assess the safety, tolerability, pharmacokinetics, and food effect of single and multiple ascending doses of ANG-3070 in healthy adult participants.

This study is comprised of 12 cohorts. 5 single ascending dose (SAD) cohorts 6multiple ascending dose (MAD) cohorts, and 1 single dose food effect (FE) cross-over cohort Each cohort will have a total of 8 subjects: SAD and MAD (2 subjects receiving placebo and 6 subjects receiving active ANG-3070)

DETAILED DESCRIPTION:
This is a Phase 1 study, to assess the safety, tolerability, pharmacokinetics, and food effect of single and multiple ascending doses of ANG-3070 in healthy adult participants.

Each cohort will have a total of 8 subjects: SAD and MAD (2 subjects receiving placebo and 6 subjects receiving active ANG-3070). The study design employs sentinel dosing with 2 subjects (1 placebo, 1 active treatment) at least 24 hours prior to remainder of cohort for dose cohort 1.

SAD cohorts are defined as follows, with the FE crossover occurring for participants in cohort A3 on Day 15 and in cohort D1 on Day 5:

A1 ANG-3070 50 mg (n=6) / Placebo (n=2) A2 ANG-3070 100 mg (n=6) / Placebo (n=2) A3 ANG-3070 200 mg (n=6) / Placebo (n=2) A3 Day 15ANG-3070 200mg (n=6) / Placebo (n=2) A4 ANG-3070 400 mg (n=6) / Placebo (n=2) A5 Day 1 ANG-3070 600 mg (n=6) / Placebo (n=2) D1 Day 1 ANG-3070 600 mg Single Dose (n=6) / Placebo (n=2) D1 Day 5 (ANG-3070 600 mg Single Dose (n=6) / Placebo (n=2)

MAD cohorts will receive drug or placebo twice daily for 14 consecutive days (Day 1 to Day 14) or drug or placebo once daily for 14 consecutive days (Day 1 to Day 14) as follows:

B1 ANG-3070 50 mg BID (n=6) / Placebo (n=2) B2 ANG-3070 100 mg BID (n=6) / Placebo (n=2) B3 ANG-3070 250 mg BID (n=6) / Placebo (n=2) B4 ANG-3070 500 mg BID (n=6) / Placebo (n=2) C1 ANG-3070 400 mg QD (n=6) / Placebo (n=2) C2 ANG-3070 600 mg QD (n=6) / Placebo (n=2)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers, aged 18 to 65 years (inclusive at the time of informed consent);
2. Participants must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of study drug; and
3. Participants must have a minimum body weight of 50 kg and a Body Mass Index (BMI) between ≥18.0 and ≤32.0 kg/m2 at Screening;

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period;
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant;
3. History of gastrointestinal (GI) disorders such as celiac disease, atrophic gastritis, lactose intolerance, and Helicobacter (H.) pylori infection;
4. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol;
5. Any surgical or medical condition that could interfere with the absorption, distribution, metabolism, or excretion of the study drug;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Difference in Adverse Events | Up to the Follow Up visit 8 days after the last study drug administration
  Difference versus placebo in the number of subjects with adverse events to evaluate safety and tolerability of ANG3070.
Difference in Vital Signs | Up to the Follow Up visit 8 days after the last study drug administration
  Difference versus placebo in the number of subjects with abnormal vital signs to evaluate safety and tolerability of ANG3070.
Difference in Physical Exam | Up to the Follow Up visit 8 days after the last study drug administration
  Difference versus placebo in the number of subjects with abnormal Physical examination to evaluate safety and tolerability of ANG3070
Difference in Lab Values | Up to the Follow Up visit 8 days after the last study drug administration
  Difference versus placebo in the number of subjects with abnormal lab values to evaluate safety and tolerability of ANG3070.
Difference in ECG QT interval | Up to the Follow Up visit 8 days after the last study drug administration
  Difference versus placebo in the number of subjects with abnormal ECG QT interval to evaluate safety and tolerability of ANG3070

SECONDARY OUTCOMES:
Assess PK | Up to the Follow Up visit 8 days after the last study drug administration
  To assess the pharmacokinetics (PK) of single and multiple ascending doses of ANG-3070 and to evaluate the effect of a high fat meal on the PK of a single dose of ANG-3070 administered to healthy adult participants

CONTACTS AND LOCATIONS:
Overall Officials: Shakil Aslam, MD, Study Director — Angion Biomedica
Locations (1):
- Nucleus Network, VIC, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Undecided